CLINICAL TRIAL: NCT05946304
Title: The Effects of Exercise Training on Physical and Mental Health in Women With Cardiac Implantable Electronic Devices (CIED-EX): a Pilot Study
Brief Title: Exercise Training in Women With Cardiac Devices
Acronym: CIED-EX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230095-01H
Record Dates: First submitted 2023-06-13; First posted 2023-07-14 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Population Groups; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care + moderate-intensity continuous exercise training (MICT) (Experimental): Supervised virtual MICT exercise sessions for 12 weeks (2x/wk) using the platform Zoom Care.
  Interventions: Behavioral: moderate-intensity continuous exercise training (MICT) group
- Standard care + high-intensity interval training (HIIT) (Experimental): Supervised virtual HIIT exercise sessions for 12 weeks (2x/wk) using the platform Zoom Care.
  Interventions: Behavioral: high-intensity interval training (HIIT) group

INTERVENTIONS:
Behavioral: moderate-intensity continuous exercise training (MICT) group — Exercise session: Warm-up: 60-70% peak heart rate (HR) - 10min; Training: 70-85% peak HR - 35min; Cool-down: 60-70% peak HR - 15min.
  Arms: Standard care + moderate-intensity continuous exercise training (MICT)
Behavioral: high-intensity interval training (HIIT) group — Warm-up: 60-70% peak heart rate (HR) - 10min; Training: 85-95% peak HR - 25 minutes (4x4-minutes of high-intensity intervals interspersed with 3 minutes of low-intensity intervals); Cool-down: 60-70% peak HR - 10min.
  Arms: Standard care + high-intensity interval training (HIIT)

SUMMARY:
Cardiac implantable electronic devices (CIED) are established treatments for a variety of cardiac arrhythmias. Women with CIED have lower fitness and lower quality of life compared to men with CIED. Moderate-intensity continuous training (MICT) is the most prescribed exercise for women. However, high-intensity interval training (HIIT) has been shown to improve fitness, anxiety levels, quality of life, and other health indicators over MICT in men with CIED. There is a need to quantitatively evaluate the feasibility and effects of a virtual HIIT vs. virtual MICT program on the physical, quality of life, and mental health of women with CIED. Furthermore, a qualitative approach is also necessary to understand patients' experiences, barriers, and facilitators of a virtual exercise intervention. This mixed-methods pilot randomized controlled trial will assess the feasibility of a 12-week virtual HIIT and MICT program in women with CIED.

ELIGIBILITY:
Inclusion Criteria:

1. Women (i.e., female sex assigned at birth) with CIED (≥6 months since implant)
2. Women with CIED in optimal medical therapy and functioning;
3. Patient is able to perform a symptom-limited CPET;
4. Patient is able to read and understand English or French.

Exclusion Criteria:

1. Patient is currently participating in routine exercise training (>2x/week);
2. Patient has: documented unstable angina; or established diagnosis of chronic obstructive pulmonary disease, severe mitral or aortic stenosis, or hypertrophic obstructive cardiomyopathy;
3. Patient has an unmanaged psychiatric illness (e.g., active psychosis, suicidal ideation) or cognitive impairment;
4. Patient does not have an internet connection or a device with a camera and speakers;
5. Patient with any device troubleshooting at resting or during exercise;
6. Patient is unable to provide written informed consent;
7. Patient is unwilling or unable to return for follow-up visits at week 12;
8. Patient is unwilling to be randomized to HIIT or MICT; or
9. Pregnancy or patients who become pregnant during the 12-week intervention phase (the effects of interval training on an unborn fetus are unknown).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Number of classes participants attended | Week 12
  Exercise attendance will be assessed by the number of classes participants attended. High attendance to the CR program will be defined as being present at ≥ 70% of the classes.
Feasibility - Compliance to the exercise prescription based on heart rate | Week 12
  Exercise compliance will be assessed as the ability to complete the prescribed intensity (based on the heart rate peak [HR] of the cardiopulmonary exercise test) for high-intensity interval training or moderate-intensity continuous training. The HRs across all classes for each patient will be averaged and compared to their target HR prescription. For instance, where patients exercised below, within, or above the prescribed HR ranges, these will be coded as "does not comply", "complies" and "exceeds".
Feasibility - Adverse events | Week 12
  Safety will be assessed by enumerating reported adverse events during the study period.
Feasibility - Number of dropouts | Week 12
  The number of patients who withdraw from the program will be reported as descriptive data and compared between groups (e.g., high-intensity interval program vs moderate-intensity continuous training).

SECONDARY OUTCOMES:
Exercise capacity - maximal oxygen uptake (VO2peak) | Baseline
  will be measured using a gold standard symptom-limited, cardiopulmonary exercise test (CPET) on an electronically braked cycle ergometer. Gas exchange will be monitored continuously; the highest rate of oxygen uptake achieved (i.e. peak VO2 in mL/kg/min) during the last minute of the CPET will represent exercise capacity.
Exercise capacity - maximal oxygen uptake (VO2peak) | Week 6
  will be measured using a gold standard symptom-limited, cardiopulmonary exercise test (CPET) on an electronically braked cycle ergometer. Gas exchange will be monitored continuously; the highest rate of oxygen uptake achieved (i.e. peak VO2 in mL/kg/min) during the last minute of the CPET will represent exercise capacity.
Exercise capacity - maximal oxygen uptake (VO2peak) | Following 12-weeks of intervention
  will be measured using a gold standard symptom-limited, cardiopulmonary exercise test (CPET) on an electronically braked cycle ergometer. Gas exchange will be monitored continuously; the highest rate of oxygen uptake achieved (i.e. peak VO2 in mL/kg/min) during the last minute of the CPET will represent exercise capacity.
Quality of life (self-reported) | Baseline
  will be measured using the 36-Item Short Form Health Survey questionnaire (SF-36). The SF-36 is a widely used and thoroughly validated, standardized, generic health survey with 36 questions. It yields an 8-scale (physical functioning; role-physical; bodily pain; general health; vitality; social functioning; role-emotional; and, mental health) profile of functional health and well-being scores as well as psychometrically-based physical (PCS) and mental (MCS) component summary scores. The PCS has been shown to be one of the most valid SF-36 scales for measuring physical health. The score ranges from 0 (low) to 100 (high). The lower the score the more disability. Higher scores indicate better health status.
Quality of life (self-reported) | Following 12-weeks of intervention
  will be measured using the 36-Item Short Form Health Survey questionnaire (SF-36). The SF-36 is a widely used and thoroughly validated, standardized, generic health survey with 36 questions. It yields an 8-scale (physical functioning; role-physical; bodily pain; general health; vitality; social functioning; role-emotional; and, mental health) profile of functional health and well-being scores as well as psychometrically-based physical (PCS) and mental (MCS) component summary scores. The PCS has been shown to be one of the most valid SF-36 scales for measuring physical health. The score ranges from 0 (low) to 100 (high). The lower the score the more disability. Higher scores indicate better health status.
Mental health - Anxiety levels | Baseline
  measured using the Generalized Anxiety Disorder 7-item (GAD-7) questionnaire.GAD-7 is a validated, self-reported anxiety questionnaire. The GAD-7 is a 7-item questionnaire developed to identify probable cases of generalized anxiety disorder. The GAD-7 score ranges from 0 - 21, where scores between 10-14 indicate moderate levels of anxiety and scores over 15 indicate severe anxiety.
Mental health - Anxiety levels | Following 12-weeks of intervention
  measured using the Generalized Anxiety Disorder 7-item (GAD-7) questionnaire.GAD-7 is a validated, self-reported anxiety questionnaire. The GAD-7 is a 7-item questionnaire developed to identify probable cases of generalized anxiety disorder. The GAD-7 score ranges from 0 - 21, where scores between 10-14 indicate moderate levels of anxiety and scores over 15 indicate severe anxiety.
Mental health - Depression levels | Baseline and following 12-weeks of intervention
  measured using the Patient Health Questionnaire (PHQ-9) questionnaire. The PHQ-9 is a nine-symptom checklist questionnaire, where each question score ranges from 0 - 3. The total score ranges from 0-27 and it is divided into 5 levels: 0-4 (minimal); 5-9 (mild); 10-14 (moderate;) 15-19 (moderately severe) and 20-27 (severe depression).
Mental health - Depression levels | Following 12-weeks of intervention
  measured using the Patient Health Questionnaire (PHQ-9) questionnaire. The PHQ-9 is a nine-symptom checklist questionnaire, where each question score ranges from 0 - 3. The total score ranges from 0-27 and it is divided into 5 levels: 0-4 (minimal); 5-9 (mild); 10-14 (moderate;) 15-19 (moderately severe) and 20-27 (severe depression).
Cardiometabolic health indicators - Blood pressure | Baseline
  Resting systolic and diastolic blood pressure will be measured in a seated position after a 5-minute rest period on the right arm using an automated, blood pressure monitor.
Cardiometabolic health indicators - Blood pressure | Following 12-weeks of intervention
  Resting systolic and diastolic blood pressure will be measured in a seated position after a 5-minute rest period on the right arm using an automated, blood pressure monitor.
Cardiometabolic health indicators - Heart rate | Baseline
  measured in a seated position after a 5-minute rest period using an automated blood pressure monitor.
Cardiometabolic health indicators - Heart rate | Following 12-weeks of intervention
  measured in a seated position after a 5-minute rest period using an automated blood pressure monitor.
Cardiometabolic health indicators - Body mass index | Baseline
  Height (cm) and body mass (kg) will be measured to compute body mass index (kg/m2).
Cardiometabolic health indicators - Body mass index | Following 12-weeks of intervention
  Height (cm) and body mass (kg) will be measured to compute body mass index (kg/m2).
Cardiometabolic health indicators - Fat mass | Baseline
  Fat mass (kg) and fat-free mass (kg) will be measured using bioelectrical impedance.
Cardiometabolic health indicators - Fat mass | Following 12-weeks of intervention
  Fat mass (kg) and fat-free mass (kg) will be measured using bioelectrical impedance.
Cardiometabolic health indicators - Waist circumference | Baseline
  will be measured using standardized procedures (2 repeated measures using a tape; in centimeters).
Cardiometabolic health indicators - Waist circumference | Following 12-weeks of intervention
  will be measured using standardized procedures (2 repeated measures using a tape; in centimeters).
Cardiometabolic health indicators - Menstrual status | Baseline
  The menstrual status will be collected via a questionnaire.
Cardiometabolic health indicators - Menstrual status | Following 12-weeks of intervention
  The menstrual status will be collected via a questionnaire.
Self-determined motivation for exercise | baseline
  the 24-item Behavioural Regulation in Exercise questionnaire (BREQ-3) yields an overall Relative Autonomy Index (RAI) score, representing overall self-determined motivation.Each item is rated on a 5-point Likert scale (0-4), with higher scores representing greater self-determined motivation for exercise.
Self-determined motivation for exercise | following 12-weeks of intervention
  the 24-item Behavioural Regulation in Exercise questionnaire (BREQ-3) yields an overall Relative Autonomy Index (RAI) score, representing overall self-determined motivation. Each item is rated on a 5-point Likert scale (0-4), with higher scores representing greater self-determined motivation for exercise.
Exercise self-efficacy | baseline
  the 9-item Multidimensional Self-Efficacy for Exercise Scale (MSES-R) yields an overall self-efficacy for exercise score reflecting scheduling, task, and coping self-efficacy. Participants are asked: "How confident are you that you can exercise when…" and respond to each item on a 100% confidence scale (0-100). A higher score indicates higher self-efficacy for exercise.
Exercise self-efficacy | following 12-weeks of intervention
  the 9-item Multidimensional Self-Efficacy for Exercise Scale (MSES-R) yields an overall self-efficacy for exercise score reflecting scheduling, task, and coping self-efficacy. Participants are asked: "How confident are you that you can exercise when…" and respond to each item on a 100% confidence scale (0-100). A higher score indicates higher self-efficacy for exercise.
Physical activity enjoyment | baseline
  the 18-item Physical Activity Enjoyment Scale (PACES) measures the extent (on a 7-point Likert scale) to which participants enjoy doing physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" from 1 (I enjoy it) to 7 (I hate it). The score ranges from 18-126. Higher scores indicate higher enjoyment.
Physical activity enjoyment | following 12-weeks of intervention
  the 18-item Physical Activity Enjoyment Scale (PACES) measures the extent (on a 7-point Likert scale) to which participants enjoy doing physical activity by asking participants to rate "how you feel at the moment about the physical activity you have been doing" from 1 (I enjoy it) to 7 (I hate it). The score ranges from 18-126. Higher scores indicate higher enjoyment.
Gender-Related Variables | baseline a
  Participants will complete the Genesis-Praxy questionnaire (20-item). The gender score is used to categorize patients according to the masculine and feminine characteristics they present (i.e., according to their gender profile). The score represents the probability between 0% and 100% for each patient to be a "woman." Therefore, the gender scale is considered a continuum, ranging from masculine characteristics (gender scores toward zero) to feminine traits (gender scores toward one hundred). This scale does not assess worse or better outcomes.
Gender-Related Variables | following 12-weeks of intervention
  Participants will complete the Genesis-Praxy questionnaire (20-item). The gender score is used to categorize patients according to the masculine and feminine characteristics they present (i.e., according to their gender profile). The score represents the probability between 0% and 100% for each patient to be a "woman." Therefore, the gender scale is considered a continuum, ranging from masculine characteristics (gender scores toward zero) to feminine traits (gender scores toward one hundred). This scale does not assess worse or better outcomes.
Gender identity | baseline
  Participants will complete the Traditional Masculinity and Femininity scale (TMF), designed to assess central facets of self-ascribed masculinity-femininity. A 7-point scale is used to gauge the extent to which the participant feels feminine or masculine (e.g., how feminine or masculine she or he ideally would like to be, and how feminine and masculine her or his appearance, interests, attitudes, and behavior would traditionally be seen). This scale does not assess worse or better outcomes.
Gender identity | following 12-weeks of intervention
  Participants will complete the Traditional Masculinity and Femininity scale (TMF), designed to assess central facets of self-ascribed masculinity-femininity. A 7-point scale is used to gauge the extent to which the participant feels feminine or masculine (e.g., how feminine or masculine she or he ideally would like to be, and how feminine and masculine her or his appearance, interests, attitudes, and behavior would traditionally be seen). This scale does not assess worse or better outcomes.

OTHER OUTCOMES:
Focus groups | Following 12-weeks of intervention
  semi-structured focus group using Zoom Healthcare with purposively selected patients to explore factors influencing compliance and satisfaction with MICT or HIIT.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Results from this study may be presented at scientific conferences and/or published in journals but participants will not be identifiable in any publications or presentations. Data can be made available upon request by contacting the principal investigator.